CLINICAL TRIAL: NCT05121675
Title: Investigating How Incentives Impact Engagement With an Online Mental Health Application (Neuroflow)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: NeuroFlow (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 849894
Record Dates: First submitted 2021-11-02; First posted 2021-11-16 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Behavioral Economics; Gifts, Financial; Point
MeSH Terms: conditions — Gift Giving

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of the two arms. The participants getting the app with behavioral economics incentives only will be enrolled at the same time as the participants getting the app with behavioral economics + financial incentives.
Who Masked: Participant
Masking Description: Participants will be randomized to one of the two groups and will not be informed of which one. If they directly ask the investigators will tell them at the end of the trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App with behavioral economics + financial incentives (Experimental): NeuroFlow uses behavioral economics reminders, gamification, and fun, motivating messages to encourage use. It also includes financial incentives so users can earn redeemable points accrued for activity completion for gift cards at popular outlets (e.g., 1000 points which is the maximum per month = $10 gift card).
  Interventions: Behavioral: Neuroflow app: Mental health and wellbeing resources for adults
- App with behavioral economics incentives only (Active Comparator): NeuroFlow uses behavioral economics reminders, gamification, and fun, motivating messages to encourage use. including points accrued for activity completion. This version of the app does not have financial incentives.
  Interventions: Behavioral: Neuroflow app: Mental health and wellbeing resources for adults

INTERVENTIONS:
Behavioral: Neuroflow app: Mental health and wellbeing resources for adults — The NeuroFlow app delivers resources on resilience training, mindfulness-based strategies and cognitive behavioral therapy to adults looking to support their mental health and wellbeing. The specific "journey" (i.e., content such as activities, videos, trackers, and journaling) is tailored to individuals based on depression and anxiety screeners administered upon signing up to the app.

SUMMARY:
The purpose of the study is to understand how incentives (either points alone or points that can be exchanged for gift certificates) encourage engagement with an online mental health app (Neuroflow) for University students. Overall, the hope of this study is to help the investigators understand how best to support mental health and wellness in university students.

DETAILED DESCRIPTION:
As mental health awareness and intervention has gained more traction throughout the years, applications - such as NeuroFlow - have emerged in an effort to facilitate aid to those who are unable to afford or access alternative mental health care methods. However, over 95% of mental health and wellness applications have not actually been studied. Additionally, a large portion examines user adoption of various mental health applications based on different factors, leaving a gap in research regarding client engagement and interest post-installation. Thus, despite promises, applications for promoting mental health often do not achieve their intended goals due to lack of sufficient client engagement/interest. In order to address this discrepancy, the use of financial incentives and other incentives from the field of behavioral economics may help. As an application, NeuroFlow embeds behavioral economic principles to increase motivation and engagement with the application (such as personalized pop-up notification reminders and app gamification including points accrual for activity completion and celebratory messages for meeting points thresholds) and also provides financial incentives whereby points accrued can be redeemed into gift cards for popular outlets such as Amazon. However, it is not clear if this financial incentive increases engagement or has knock-on effects for mental health and wellbeing over and above the behavioral economics incentives per se. In this study, the investigators will conduct a pilot two-arm randomized controlled trial where the investigators will examine the effect of a treatment group (NeuroFlow app with behavioral economics and financial incentives vs. NeuroFlow app with behavioral economics incentives only) on application engagement and mental health and wellbeing (anxiety and depression symptoms, sleep, self-regulation and wellbeing). The purpose of this study is to gain an understanding of how incentives encourage participation and engagement with an online mental health platform, NeuroFlow.

This study is a two-arm pilot randomized controlled trial to assess differences in user retention and usage rates associated with two incentive structures within the NeuroFlow app (I.e., general structure versus financial compensation). The investigators will assess user engagement with utilization data (ie., daily, weekly, and monthly active users) and measures of the total number of activity counts completed by a user. After consenting to participate in the study, participants will be randomly assigned to use Neuroflow either with points only or with points and the opportunity to exchange those points for gift cards. In both conditions, participants will begin by completing a consent form and a brief questionnaire with their contact information, which will be used to grant them access to the Neuroflow platform.

In both recruitment methods, participants will be required to sign up for a 15 minute check in and check out meeting before and after the trial to answer participant questions regarding the app/app set up or concerns about the consent form. Furthermore, a Qualtrics survey will also be dispersed to participants to be taken during this time along with an initial baseline assessment (to be administered in the NeuroFlow app).

Baseline and post-app usage Qualtrics survey links will also be sent with measures (Generalized anxiety disorder (GAD), Patient Health Questionnaire (PHQ), World Health Organization- Five Well-Being Index (WHO-5), and Difficulties in Emotion Regulation Scale (DERS)) to participants in order to assess differences in user retention.

In both conditions, participants will use the Neuroflow app throughout the duration of the 4-week study (28 days). Participants will be sent a push notification each day through the app to complete their daily activities, which could include surveys, videos, or skill-based practice materials.

With the collaboration of the Neuroflow team, the usage metrics of the app will be pulled after the end of the study. The user metrics of interest are identifying factors that include first name, last name, gender, age, date of birth, and the applicable assignments to each participant - care team manager and behavioral health specialist. Additionally, the first and last score, first and last date, and time between the first and last assessment dates for the measures of interest (PHQ-9, GAD-7, WHO-5, DERS). Furthermore, the total activity number and the total activity rate across all measures will be collected. No additional data from or about participant phone usage or activities will be pulled as part of the study other than the usage metrics specified above, specific to Neuroflow.

ELIGIBILITY:
Inclusion Criteria:

* The target population for this study are college students either at the University of Pennsylvania or other US universities. Participants will be included if they have a smartphone and are willing to download and use the Neuroflow app throughout the duration of the study

Exclusion Criteria:

* Does not own a smartphone capable of downloading the NeuroFlow application or is unwilling to download and use the Neuroflow app throughout the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Nuske, Principal Investigator — Penn Medicine
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang HY, Bashir M. Users' Adoption of Mental Health Apps: Examining the Impact of Information Cues. JMIR Mhealth Uhealth. 2017 Jun 28;5(6):e83. doi: 10.2196/mhealth.6827. PMID 28659256
- [Background] Huckvale K, Nicholas J, Torous J, Larsen ME. Smartphone apps for the treatment of mental health conditions: status and considerations. Curr Opin Psychol. 2020 Dec;36:65-70. doi: 10.1016/j.copsyc.2020.04.008. Epub 2020 May 4. PMID 32553848
- [Background] Lecomte T, Potvin S, Corbiere M, Guay S, Samson C, Cloutier B, Francoeur A, Pennou A, Khazaal Y. Mobile Apps for Mental Health Issues: Meta-Review of Meta-Analyses. JMIR Mhealth Uhealth. 2020 May 29;8(5):e17458. doi: 10.2196/17458. PMID 32348289

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants were college students at the University of Pennsylvania who had access to a smartphone and agreed to download and use the NeuroFlow application
Period: Overall Study
Arm/Group | App With Behavioral Economics + Financial Incentives | App With Behavioral Economics Incentives Only
Started | 53 | 54
Completed | 48 | 39
Not Completed | 5 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | App With Behavioral Economics + Financial Incentives | App With Behavioral Economics Incentives Only | Total
Number analyzed (Participants) | 53 | 54 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 54 | 107
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.7 (1.8) | 19.4 (1.1) | 19.5 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: some did not report gender
  Participants
    number analyzed (Participants) | 41 | 44 | 85
    Female | 23 | 29 | 52
    Male | 18 | 15 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 15 | 30
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 4 | 10
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 16 | 28
Region of Enrollment [Number; unit: participants]
  United States | 53 | 54 | 107

OUTCOME MEASURES:

1. Primary Outcome: Engagement (Percentage of Daily check-in Activities)
Description: User engagement will be measured as the percentage of daily check-in activities (number completed out of the total number of activities assigned)
Time Frame: Throughout 28-day trial (averaged)
Population: some dropped out
Measure: Mean (Standard Error); unit: percentage of completion
Arm/Group | App With Behavioral Economics + Financial Incentives | App With Behavioral Economics Incentives Only
Number analyzed (Participants) | 48 | 39
percentage of completion | 32.8176 (2.89863) | 30.242 (3.18953)

2. Secondary Outcome: Generalized Anxiety Disorder (GAD-7)
Description: Change from pre-trial to post-trial score in anxiety. Scores range from 0 to 21. Higher scores = higher symptoms of anxiety.
Time Frame: Baseline and post-trial, up to 28 days
Population: some dropped out
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | App With Behavioral Economics + Financial Incentives | App With Behavioral Economics Incentives Only
Number analyzed (Participants) | 27 | 34
score on a scale
  Baseline | 6.58 (0.781) | 6.71 (0.653)
  Post Trial | 4.45 (0.692) | 5.19 (0.779)

3. Secondary Outcome: Patient Health Questionnaire (PHQ-8)
Description: Change from pre-trial to post-trial score in depression. Scores range from 0-24. Higher scores = higher symptoms of depression.
Time Frame: Baseline and post-trial, up to 28 days
Population: some dropped out
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | App With Behavioral Economics + Financial Incentives | App With Behavioral Economics Incentives Only
Number analyzed (Participants) | 31 | 41
score on a scale
  Baseline | 5.45 (0.365) | 6.08 (0.374)
  Post Trial | 4.62 (0.434) | 5.3 (0.427)

4. Secondary Outcome: World Health Organization (WHO-5)
Description: Change from pre-trial to post-trial score in wellbeing. Scores range from 0-100 (raw score is multiplied by 4). Higher scores = higher wellbeing.
Time Frame: Baseline and post-trial, up to 28 days
Population: some dropped out
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | App With Behavioral Economics + Financial Incentives | App With Behavioral Economics Incentives Only
Number analyzed (Participants) | 33 | 41
score on a scale
  Baseline | 57.95 (0.361) | 55.9 (0.369)
  Post Trail | 58.89 (0.393) | 61.45 (0.409)

5. Secondary Outcome: Difficulties Emotion Regulation Scale (DERS)
Description: Change from pre-trial to post-trial score in emotion regulation difficulties. Scores range from 36-180. Higher scores = greater problems with emotion regulation.
Time Frame: Baseline and post-trial, up to 28 days
Population: some dropped out
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | App With Behavioral Economics + Financial Incentives | App With Behavioral Economics Incentives Only
Number analyzed (Participants) | 31 | 41
score on a scale
  Baseline | 83.29 (0.365) | 83.22 (0.369)
  Post Trail | 76.36 (0.409) | 74.32 (0.421)

ADVERSE EVENTS:
Time Frame: 1 month
Description: Adverse events were assessed during the post-trial interviews for all participants. Additionally, any participant logs in the NeuroFlow app that included descriptions of self-harm were flagged.
Arm/Group | App With Behavioral Economics + Financial Incentives | App With Behavioral Economics Incentives Only
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/54
Other Adverse Events (participants affected / at risk) | 0/53 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT05121675/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT05121675/ICF_001.pdf